CLINICAL TRIAL: NCT00572143
Title: Should the Surgeon or the General Practitioner (GP) Follow up Patients After Surgery for Colon Cancer? A Randomized Controlled Trial Focusing on Quality of Life, Cost-effectiveness and Serious Clinical Events.
Brief Title: Follow-up After Surgery for Colon Cancer. General Practice vs. Surgical-based Follow-up?
Acronym: ONKOLINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P-REK NORD 79/2006
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Colon Cancer
Keywords: Colonic Neoplasms/surgery*; Continuity of Patient Care*; Follow-Up Studies; Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Colonic Neoplasms; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Postoperative follow-up of ca coli patients at the surgical outpatient dpt
  Interventions: Other: ca coli follow-up by GP
- 2 (Active Comparator): Postoperative follow-up of ca coli patients by GP's
  Interventions: Other: ca coli follow-up by GP

INTERVENTIONS:
Other: ca coli follow-up by GP — patients randomized to follow up by GP

SUMMARY:
The purpose of this study is to clarify cost effectiveness and quality of life issues among colon cancer patients followed up in a hospital setting or by their GP's.Statement of study hypothesis:Postoperative follow up of colon cancer patients (according to national guidelines) by general practitioners will not have any influence on patients' quality of life. There will not be observed any increase in serious clinical events and cost effectiveness will be improved.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for colon cancer (including rectosigmoid) with histological grade Duke stages A, B or C.
* Completion of postsurgical chemotherapy (Dukes stage C patients).
* Informed consent.

Exclusion Criteria:

* Patients with rectal cancer defined as cancer within 15 cm from anus.
* A poor health status or operative complications making it natural to perform follow up by specialists.
* Additional cancer diagnoses.
* Disseminated cancer.
* Poor mental status.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quality of life; EORTC-QLQ-C30 and EQ 5D | 2 years

SECONDARY OUTCOMES:
Cost-effectiveness Serious clinical events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rolv-Ole Lindsetmo, MD, PHd, Study Chair — University of Tromso; Caroline Sagatun, MD, Principal Investigator — Bodø Hospital Trust; Niels Krum-Hansen, Principal Investigator — University Hospital of North Norway (Harstad)
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Augestad KM, Norum J, Rose J, Lindsetmo RO. A prospective analysis of false positive events in a National Colon Cancer Surveillance Program. BMC Health Serv Res. 2014 Mar 27;14:137. doi: 10.1186/1472-6963-14-137. PMID 24674307
- [Derived] Augestad KM, Norum J, Dehof S, Aspevik R, Ringberg U, Nestvold T, Vonen B, Skrovseth SO, Lindsetmo RO. Cost-effectiveness and quality of life in surgeon versus general practitioner-organised colon cancer surveillance: a randomised controlled trial. BMJ Open. 2013 Apr 4;3(4):e002391. doi: 10.1136/bmjopen-2012-002391. Print 2013. PMID 23564936
- [Derived] Augestad KM, Vonen B, Aspevik R, Nestvold T, Ringberg U, Johnsen R, Norum J, Lindsetmo RO. Should the surgeon or the general practitioner (GP) follow up patients after surgery for colon cancer? A randomized controlled trial protocol focusing on quality of life, cost-effectiveness and serious clinical events. BMC Health Serv Res. 2008 Jun 25;8:137. doi: 10.1186/1472-6963-8-137. PMID 18578856